CLINICAL TRIAL: NCT00156780
Title: A Phase 1, Double Blind, Crossover, Placebo-Controlled, Dual-Injection, Safety and Pharmacokinetic Study of AI-700 in Patients With Diminished DLCO and Chronic Obstructive Pulmonary Disease (COPD) and/or Congestive Heart Failure (CHF)
Brief Title: Phase 1 Safety and Pharmacokinetic Study of AI-700 in Patients With Diminished DLCO and COPD and/or CHF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acusphere (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: AI-700-05
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-07

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: ultrasound contrast agent; pharmacokinetics; congestive heart failure; chronic obstructive pulmonary disease; safety
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — perfluorobutane

INTERVENTIONS:
Drug: AI-700

SUMMARY:
This study was conducted to evaluate the safety and pharmacokinetics of an echocardiographic contrast agent, AI-700, in patients with moderate to severe chronic obstructive pulmonary disease (COPD) and/or congestive heart failure (CHF).

DETAILED DESCRIPTION:
In ongoing clinical trials, AI-700 is currently being evaluated for its value to provide enhanced echocardiography to detect CAD. The patient population is comprised of those patients who have chest pain and are being evaluated for inducible ischemia. This population may include patients with compromised pulmonary function due to COPD or CHF. This study was to evaluate the safety of AI-700 in these patients.

Age Groups: Child, Adult, Older Adult
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
To determine the safety of AI-700 in patients with diminished pulmonary diffusing capacity (DLCO) and moderate or severe COPD and/or CHF
To determine the pharmacokinetics of perfluorocarbon gas in blood following an intravenous injection of AI-700 in this patient population

CONTACTS AND LOCATIONS:
Locations (1):
- Acusphere, Inc., Watertown, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.acusphere.com